CLINICAL TRIAL: NCT05585372
Title: EFFECT OF RADIOLOGICAL GUIDED MOBILIZATION ON CERVICAL INTERVERTEBRAL FORAMEN IN PATIENTS WITH CANAL STENOSIS
Brief Title: EFFECT OF CT GUIDED MOBILIZATION ON CERVICAL FOREMAN'S DIMENSIONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Aly, Mahmoud Mohamed Aly, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT guided C Sp F Mobilization.
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: EFFECT OF CT Guided Mobilization ON CERVICAL RADICULOPATHY

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The control group will receive general stability exercises and neurodynamic mobilization only
- CT guided opening mobilization of cervical intervertebral foreman (Experimental): Grade four manual therapy mobilization of cervical intervertebral foreman guided by 3 dimensions computed tomography (CT) as following :
  1. Determining the poper direction of cervical IVF by 3D CT.
  2. the patients lies in supine with his head resting comfortably at the position which cause maximum opening of the intervertebral foramen which has been determined by the 3D CT.
  3. cervical lateral glide from right to left for C5, C6 and C7, Grade IV 3 × 6 on each segment.
  4. Passive mobilization techniques were progressed, utilizing unilateral posteroanterior mobilization of the mid and lower cervical spine and lateral gliding movements, in both directions, progressing in duration and intensity to allow a graded exposure of load.
  5. Sustained Natural Apophyseal Glides (SNAGS) were used mainly as self-treatment techniques to maintain the gains that achieved.
  Interventions: Other: CT guided opening mobilization of cervical intervertebral foreman

INTERVENTIONS:
Other: CT guided opening mobilization of cervical intervertebral foreman — 1. the patients lies in supine with his head resting comfortably at the position which cause maximum opening of the intervertebral foramen which has been determined by the 3D CT.
  2. cervical lateral glide from right to left for C5, C6 and C7, Grade IV 3 × 6 on each segment.
  3. Passive mobilization techniques were progressed, utilizing unilateral posteroanterior mobilization of the mid and lower cervical spine and lateral gliding movements, in both directions, progressing in duration and intensity to allow a graded exposure of load.
  4. Sustained Natural Apophyseal Glides (SNAGS) were used mainly as self-treatment techniques to maintain the gains that achieved.
  Arms: CT guided opening mobilization of cervical intervertebral foreman

SUMMARY:
Applying specific opening mobilization of cervical intervertebral foramen is still unclear as well as the effect of mobilization on intervertebral foramen dimensions. using CT guidance to determine the wright direction of mobilization through studying the kinematics of intervertebral foramen will enhance better results and less risk of mobilization during manual therapy of cervical canal stenosis.

DETAILED DESCRIPTION:
The purpose of the present study is:

1. To measure dimensions of cervical intervertebral foramen in case of peripheral canal stenosis
2. To study the effect of uniaxial positions and multi axial positions on the dimensions of intervertebral foramen in case of cervical foraminal stenosis
3. To detect the proper direction of opening mobilization for cervical intervertebral foramen
4. To test the effect of applying grade four Maitland mobilization to the affected spinal unit IVF.
5. To study the effect mobilization on the cervical intervertebral foramen OF C5/6.
6. To study the effect of specific mobilization on the cervical radiculopathy

subjects and methods:

1. Thirty male patients represent the sample of this study.
2. The age of the patients range from 25 to 40 years. The body weight range from 75 to 90kg. The height range from 175 to 185Cm.
3. Each patient has disc prolapse at C5-C6 and the duration of illness ranged from three months to one year.
4. Each patient suffers from cervical radiculopathy from disc prolapse at C5-C6 and the duration of illness range from three months to one year.
5. Each patient will be subjected to physical, neurological examination (motor assessment, sensory assessment) and electrophysiological assessment (H-reflex).
6. Each patient will be subjected to 3D CT scan from 6 separate positions in two visits to the Alpha Scan Radiology lab, 3 positions in each visit to avoid over dose of exposure to X ray.
7. The six positions are:

   * Neutral
   * Side bending
   * Axial rotation
   * Flexion with ipsilateral rotation
   * Flexion with contralateral
   * Extension with contralateral rotation
8. IVF width & Hight will be measured from the 3D CT from each position for Right (Rt) & left (Lt) IVF.
9. Direction of CT scan volume will 45 degree with sagittal plan and 10 to 15 degrees below the transverse plane.

Limitations:

An effort will be made to minimize the effect of the possible errors. The limitations of the study are mostly due to:

* Difference of psychological status of the patients.
* Cost of Radiological imaging processing.
* Time consuming.

Basic assumption:

It will be assumed that:

1. The psychological and environmental aspects are the same for all subjects during the study.
2. Every subject will exert the maximum effort during the study.

Null hypothesis:

1. There is no significant difference in C5-6 IVF width and height among each one of the 6 positions that Will be scanned by the 3DCT.
2. There is no significant difference in pre & post 3 months measurements of C5-6 IVF width and height in neutral positions that will be measured by the 3DCT.

ELIGIBILITY:
Inclusion Criteria:

1. All patients suffer from paramedian cervical disc prolapse (C5-C6) for at least three months up to one year. The age of the patient range from 25 to 40 years. The body weight range from 75 to 90kg. The height ranged from 175 to 185cm.
2. All the patients has unilateral cervical radiculopathy.
3. Diagnosis will be confirmed by clinical and radiological assessment (CT or MRI).

Exclusion Criteria:

* 1. Sever central canal stenosis and cervical myelopathy . 2. Sequestrated and migrated disc prolapse. 3. Acute onset of pain (pain less than three months). 4. Presence of active infection in cervical spine. 5. Postoperative cases. 6. Patient suspected to chemotherapy and radiotherapy. 7. Cervical instability.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Dimension of cervical intervertebral foreman. | 3 months
  Width and Height of Cervical intervertebral foreman measured by 3 Dimensions Computed Tomography (CT.)

SECONDARY OUTCOMES:
Neck Disability index (NDI) | 6 weeks
  Neck pain and function Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sameha H Hassan, professor, Study Chair — professor of physical therapy for neuromuscular disorders and its surgery
Locations (1):
- ElRazzy Spine physical therapy clinics, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided